CLINICAL TRIAL: NCT05478876
Title: CNAO 40-2020 C CYCLE "Carbon Ion Radiation Therapy in the Treatment of Mucous Melanomas of the Female Lower Genital Tract" "Radioterapia Con Ioni Carbonio Per il Trattamento Dei Melanomi Mucosi Ginecologici"
Brief Title: Carbon Ion Radiation Therapy in the Treatment of Mucous Melanomas of the Female Lower Genital Tract
Acronym: CYCLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNAO 40-2020 C CYCLE
Record Dates: First submitted 2021-12-29; First posted 2022-07-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Malignant Melanoma; Gynecologic Cancer
Keywords: hadrontherapy, gynecological melanoma
MeSH Terms: conditions — Melanoma | interventions — Heavy Ion Radiotherapy; Immunotherapy

STUDY DESIGN:
Intervention Model Description: cohort of 9 patients with primary gynecological melanoma. The intervention consists in carbon ion radiation therapy.
  The expected duration of treatment is 4 weeks, 4 fractions per week.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- carbon ion radiotherapy (Experimental): Patients affected by pelvic recurrence of gynecological cancer, who had not undergone to previous pelvic irradiation, will be enrolled on this study. After enrollment, patients undergo baseline exams, simulation CT and MRI and then carbon ion radiation therapy treatment will be performed, according to trial indications.
  Interventions: Radiation: carbon ion radiation therapy CIRT

INTERVENTIONS:
Radiation: carbon ion radiation therapy CIRT — CIRT: The low-dose CTV (clinical target volume) will receive a total dose of 43 GyRBE in 10 fractions, 4 fractions per week. The high-dose CTV will receive a total dose of 68.8 GyRBE in 16 fractions, 4 fractions per week.
  The expected duration of treatment is 4 weeks, 4 fractions per week. Treatments lasting longer than 6 weeks, or with less than 6 fractions administered on 14 consecutive days, will not be considered acceptable.
  Immunotherapy: Patients will undergo immunotherapy after carbon ion radiation therapy (CIRT) up to maximum response and/or up to tolerance. The concomitant association of immunotherapy is not envisaged in this protocol.
  Other Names: immunotherapy

SUMMARY:
The present monocentric prospective phase 2 study aims to reproduce the results obtained at NIRS thus offering the possibility of obtaining a promising rate of progression-free survival (PFS) and local control (LC) in patients diagnosed with mucosal melanoma of lower genital tract. Systemic treatment with immunotherapy is not the subject of this study but is allowed both in the neoadjuvant and sequential regimens.

Melanomas have always been considered poorly radiosensitive. It is now accepted that high LET (Linear Energy Transfer) particle beams, such as carbon ions, can offer a biological advantage, compared to photons treatment, in radio-resistant neoplasms treatment, thanks to their higher biological efficacy (RBE) against tumours with a low α/ ß ratio. In addition, carbon ions have the physical advantage of an inverted depth deposition profile compared to photons, allowing then a steep dose gradients that ensure increased sparing of adjacent healthy organs at risk (OARs).

DETAILED DESCRIPTION:
Patients with primary gynaecological melanoma, non-metastatic, non-suitable for surgery, and not previously subjected to conventional radiotherapy can be enrolled in the trial, according to selection criteria. After requested baseline exams, the patient undergoes to simulation phase for the carbon ion radiation therapy, according to study constraints. The patient will then receive immunotherapy not concomitant to CIRT. The response is evaluated through RECIST criteria.

PFS is the primary endpoint, calculated from the end of CIRT to date of disease progression or death or last follow up.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis
* Absence of skin extension
* N + (only if confined to the groin and pelvis)
* Age between 20-80 years
* ECOG 0-2
* No evidence of metastasis
* At least 5 mm away with rectum and bladder wall
* No previous RT
* Written informed consent
* Patient's ability to understand the characteristics and consequences of the clinical trial
* Molecular characterization/ mutational state
* Disease staging (baseline exams)

Exclusion Criteria:

* Hip prosthesis, or metal prostheses or any other condition that prevents adequate imaging to identify the target volume and calculate the dose in the treatment plan
* Psychic or other disorders that may prevent informed consent
* Previous invasive tumor unless patient has been disease free for at least 3 years
* Contraindication to MRI
* Pregnancy or breastfeeding in progress

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gynecological disease
Enrollment: 9 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 years
  estimate 2-year PFS in patients diagnosed with mucosal melanoma of the lower genital tract, treated with carbon ion radiation therapy.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  The OS will be calculated from the end date of therapy with carbon ion radiation
Toxicity according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0) | within 3 months, 3-6 months, over 6 months from CIRT
  acute, medium term and late toxicity
local response | 3 years
  according to Response Evaluation Criteria in Solid Tumours RECIST 1.1
assessment of quality of life | 3 years
  assessed through questionarie Portec 3 administered on each follow up
assessment of quality of life for >= 75 years old patients | 3 years
  assessed through questionnaire G8 Geriatric questionnaire administered on each follow up

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Barcellini, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Italy